CLINICAL TRIAL: NCT06721741
Title: Clinical and Radiographic Success of Nusmile Bioflex Versus Stainless-Steel Crowns in Restoring Decayed Primary Molars with Modified Hall Technique:A Randomized Clinical Study
Brief Title: Clinical and Radiographic Success of Nusmile Bioflex Versus Stainless-Steel Crowns in Restoring Decayed Primary Molars with Modified Hall Technique
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, hajer ahmed mousa mohamed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bioflex crowns
Record Dates: First submitted 2024-10-02; First posted 2024-12-06 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-11

CONDITIONS: Restoration of Primary Molars with Bioflex Crowns

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stainless steel crown (Active Comparator): Control group
  Interventions: Other: Stainless steel crowns
- Bioflex crown (Experimental): Intervention group
  Interventions: Other: Nusmile bioflex crowns

INTERVENTIONS:
Other: Nusmile bioflex crowns — The Bioflex crown is a new synthetic crown that has been introduced in pediatric practice. This crown is believed to offer better adaptation, durability, and ease of handling, along with improved aesthetic properties when compared to conventional crowns
  Arms: Bioflex crown
Other: Stainless steel crowns — Preformed metal crowns are a popular and affordable option as a treatment for dental caries. They offer full crown coverage and help to prevent recurrent caries. However, their aesthetic limitation is a notable drawback
  Arms: Stainless steel crown

SUMMARY:
This pilot study aims to compare the clinical and radiographic success of Bioflex (Nusmile) crowns Versus Stainless-steel crowns in restoring decayed primary molars.

DETAILED DESCRIPTION:
Decayed primary teeth must be treated promptly because they are crucial for chewing, speaking, and holding the space for permanent teeth. Losing primary teeth too early can cause various issues, including psychological problems. Hence, restoring decayed primary teeth is an essential aspect of pediatric dentistry Preformed metal crowns are a popular and affordable option as a treatment for dental caries. They offer full crown coverage and help to prevent recurrent caries. However, their aesthetic limitation is a notable drawback Parents are increasingly concerned about the appearance of dental restorations for their children and prefer tooth-colored options. To overcome this issue, Nusmile has introduced a new type of crown called "Bioflex". These crowns combine the best qualities of both stainless steel and zirconia crowns, as they are flexible, adaptable, and durable

ELIGIBILITY:
Inclusion Criteria:

* Clinical Criteria:

  1. Children from age 4-7.
  2. Cooperative children and willing for follow-up visits.
  3. Mandibular second Primary molars with multi-surface caries
* Radiographic criteria:

  1. Mandibular second Primary molars with at least two-thirds of the root remaining.

     Exclusion Criteria:
     * • General Criteria:

  <!-- -->

  1. •Unable to attend follow-up visits
  2. •Refuse to participate in the study
  3. •Uncooperative child
* Clinical Criteria:

  1. • Tooth with grade II or grade III mobility
  2. •Children with bruxism
  3. • Pulpally involved teeth
* Radiographic Criteria:

  1. •Tooth with pathological root resorption
  2. •Teeth with root caries

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Patient relevant criteria | 1 Year
  1. Clinically Success if:
     No clinical signs or symptoms like:
     * Pain
     * Dental Abscess/Swelling
     * Sinus Tract/ Fistula
     * Mobility
  2. Radiographically Success if:
  No pathology visible on x-ray like:
  * Internal/External Root Resorption
  * Peri-radicular Radiolucency
  * Furcation Involvement
  * Periapical Pathosis

SECONDARY OUTCOMES:
Crown Relevant Criteria | 1Year
  • wear of the opposing Binary (yes or no)

IPD SHARING:
Plan to Share IPD: No